CLINICAL TRIAL: NCT03833895
Title: The Phenylephrine vs. Norepinephrine Infusion by Lidico Monitoring With Pregnancy Patients Undergoing Cesarean Section
Brief Title: The Phenylephrine vs. Norepinephrine Infusion Undergoing Cesarean Section
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: China International Neuroscience Institution (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CINI-AD-201812-3
Record Dates: First submitted 2019-01-20; First posted 2019-02-07 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Cesarean Section Complications
Keywords: Cesarean delivery
MeSH Terms: interventions — Norepinephrine; Metals, Alkali; Phenylephrine; Metals, Alkaline Earth; Ringer's Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 Elements (Experimental): Continuously infusion of 0.05ug/kg/min Norepinephrine during the Cesarean Section operation
  Interventions: Drug: Norepinephrine
- Group 2 Elements (Experimental): Continuously infusion of 0.25ug/kg/min phenylephrine during the Cesarean Section operation
  Interventions: Drug: Phenylephrine
- Group 3 Elements (Placebo Comparator): In the placebo-control group, 3 ml/kg/min of LR was administrated according to standard weight.
  Interventions: Drug: Ringer's Solution

INTERVENTIONS:
Drug: Norepinephrine — 0.05ug/kg/min Norepinephrine during Cesarean Section Operation
  Other Names: Group 1 Elements
  Arms: Group 1 Elements
Drug: Phenylephrine — 0.25ug/kg/min phenylephrine during Cesarean Section Operation
  Other Names: Group 2 Elements
  Arms: Group 2 Elements
Drug: Ringer's Solution — 3 ml/kg/min of LR was administrated according to standard weight.
  Other Names: Group 3 Elements
  Arms: Group 3 Elements

SUMMARY:
Compare 0.05 μg/kg/min Norepinephrine and 0.25 μg/kg/min phenylephrine effect on fetus and parturient during Cesarean Section

DETAILED DESCRIPTION:
1. Compare 0.05 μg/kg/min Norepinephrine and 0.25 μg/kg/min phenylephrine and control group effect on parturient hemodynamic change (systolic blood pressure SBP, diastolic blood pressure DBP,mean arterial pressure MAP,heart rate HR) and on LIDICO-rapid monitoring ( stroke volume SV, systemic vascular resistance SVR, cardiac output CO) and peripheral vein (PV) blood gas during Cesarean Section.
2. Compare 0.05 μg/kg/min Norepinephrine and 0.25 μg/kg/min phenylephrine and control group effect on fetus by blood gas of the umbilical vein (UV), umbilical artery (UA),

ELIGIBILITY:
Inclusion Criteria:

* a healthy singleton pregnancy scheduled for elective cesarean delivery (CD) under combined spinal-epidural anesthesia (CSEA),
* American Society of Anesthesiologists (ASA) physical status I/II
* 20 to 40 years old

Exclusion Criteria:

* history of mental disorder or epilepsy,
* tricyclic or imipramine antidepressant use,
* central nervous system (CNS) disease,
* preexisting or pregnancy-induced hypertension,
* lumbar injury,
* severe hypovolemia,
* allergy
* history of hypersensitivity to vasopressor
* body mass index (BMI) >40 kg/m2,
* infection at the puncture site

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 238 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-02 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure (SBP) change as the one of hemodynamic outcome in general monitoring | through study completion, an average of 24 hour
  Systolic blood pressure (SBP)
Diastolic blood pressure (DBP) change as the one of hemodynamic outcome in general monitoring | Through study completion
  Diastolic blood pressure (DBP)
Mean arterial pressure (MAP) change as the one of hemodynamic outcome in general monitoring | An average of 24 hour
  Mean arterial pressure (MAP)
Heart rate (HR) change as the one of hemodynamic outcome in general monitoring | Through the study completion, an average of 24 hour
  Heart rate (HR)
Stroke volume (SV) as the part of LIDICO-rapid monitoring parameter for parturient | Through study completion, an average of 24 hour
  Stroke volume (SV)
Cardiac output (CO) as the part of LIDICO-rapid monitoring parameter for parturient | Through study completion, an average of 24 hour
  Cardiac output (CO)
Systemic vascular resistance (SVR) as the part of LIDICO-rapid monitoring parameter for parturient | Through study completion, an average of 24 hour
  Systemic vascular resistance (SVR)

SECONDARY OUTCOMES:
The benefits to the fetus based on umbilical vein (UV) blood gas | Through study completion, an average of 24 hour
  The umbilical vein (UV) blood gas
The benefits to the fetus based on umbilical artery (UA) blood gas | Through study completion, an average of 24 hour
  The umbilical artery (UA) blood gas
The benefits to parturient based on peripheral vein (PV) blood gas | Through study completion, an average of 24 hour
  Peripheral vein (PV) blood gas

CONTACTS AND LOCATIONS:
Overall Officials: Tianlong Wang, MD,PHD, Study Chair — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feng K, Wang X, Feng X, Zhang J, Xiao W, Wang F, Zhou Q, Wang T. Effects of continuous infusion of phenylephrine vs. norepinephrine on parturients and fetuses under LiDCOrapid monitoring: a randomized, double-blind, placebo-controlled study. BMC Anesthesiol. 2020 Sep 7;20(1):229. doi: 10.1186/s12871-020-01145-0. PMID 32894044